CLINICAL TRIAL: NCT01989780
Title: Bevacizumab Plus Paclitaxel Optimization Study With Interventional Maintenance Endocrine Therapy in Advanced or Metastatic ER-positive HER2-negative Breast Cancer -BOOSTER Trial, a Multicenter Randomized Phase II Study-
Brief Title: Bevacizumab Plus Paclitaxel Optimization Study With Interventional Aintenance Endocrine Therapy in Breast Cancer
Acronym: BOOSTER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Breast Cancer Research Group (Other)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JBCRG-M04; UMIN000012179 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-11-04; First posted 2013-11-21 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Bevacizumab; Letrozole; Anastrozole; exemestane; Fulvestrant; Goserelin; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): weekly paclitaxel + bevacizumab
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab
- Arm B (Experimental): endocrine therapy* + bevacizumab then back to weekly paclitaxel + bevacizumab therapy
  (*Letrozole, Anastrozole, Exemestane, Fulvestrant, LHRH Analogs + Aromatase inhibitors.)
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab; Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Goserelin; Drug: leuprorelin

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
Drug: Bevacizumab
  Other Names: Avastin
Drug: Letrozole
  Other Names: Femara
  Arms: Arm B
Drug: Anastrozole
  Other Names: Arimidex
  Arms: Arm B
Drug: Exemestane
  Other Names: Aromasin
  Arms: Arm B
Drug: Fulvestrant
  Other Names: Faslodex
  Arms: Arm B
Drug: Goserelin
  Other Names: Zoladex
  Arms: Arm B
Drug: leuprorelin
  Other Names: Leuplin
  Arms: Arm B

SUMMARY:
To compare continuing bevacizumab + paclitaxel or switching to bevacizumab + endocrine maintenance therapy followed by bevacizumab + paclitaxel, after 1st line induction therapy with bevacizumab + paclitaxel in ER+HER2- advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
This multicenter, randomized Phase II study of patients with advanced or metastatic estrogen receptor-positive human epidermal receptor type 2-negative breast cancer aims to compare two treatment strategies following induction therapy with 4-6 cycles of the combined use of weekly paclitaxel (wPTX) and bevacizumab (BV). In arm A, wPTX+BV is continued, while in arm B, wPTX is switched to maintenance endocrine therapy (hormone+BV) until disease progression, followed by wPTX+BV re-induction. The primary endpoint is time to failure of strategy, which is the time from randomization to a qualifying event (addition of a new agent not in the primary regimen, progressive disease during or after planned therapy, or death).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the breast
2. Female aged 20-75 years old at getting informed consent
3. HER2 negative disease (IHC 0/1+ or 2+ with FISH negative)
4. Documented estrogen receptor (ER) positive (>=1% by IHC)
5. Inoperative locally advanced or metastatic breast cancer at enrolment
6. Performance status (ECOG): 0-1 at enrolment
7. Life expectancy of at least 3 months from enrolment
8. No prior systemic therapy for recurrent breast cancer (excluding hormone therapy)
9. No prior neo and/or adjuvant chemotherapy with taxane or adjuvant setting with a disease-free interval from completion of the taxane treatment to metastatic diagnosis of >= 12 months
10. Patients with measurable lesion regarding with Response Evaluation Criteria in Solid Tumors(RECIST) criteria or who have evaluable lesion
11. Patients with only bone lesion will be acceptable if the osteolytic lesion has a measurable soft tissue component by MRI or CT
12. No influence on protocol treatment is considered in case prior therapy or examination.
13. Adequate following organ function within 2 weeks before starting treatment. The latest examination results should be adopted and blood transfusion or treatment of hematopoietic factor drugs is not allowed 2 weeks before examination.

    * Absolute neutrophil count >= 1500 /mm3 or white blood cell(WBC) count >= 3000 /mm3
    * Platelets >=10 x 10000 /mm3
    * Hb >= 9 g/dL
    * Total bilirubin <= 1.5 mg/dL
    * aspartate aminotransferase(AST) and alanine aminotransferase(ALT) <= 100 international unit(IU)/L
    * Serum creatinine <= 1.5 mg/dL
    * Urine dipstick for proteinuria <= 1+
14. Written informed consent signed by patients before completing any treatment related procedure

Exclusion Criteria:

1. Prior therapy with bevacizumab
2. Active infection requiring intrvenous antibiotics at enrollment or infection with active HBV and/or HCV.
3. Pregnancy, lactetion or in case of potentialy pregnancy women Not mind contraception in trial period.
4. Known hypersensitivity to bevacizumab or paclitaxel
5. History of hemoptysis (>= 2.5mL of bright red blood per episord).
6. Use of disulfiram,cyanamide, carmofur or procarbazine Hydrochloride
7. Patients with CNS metastases (except for not symptomatic)
8. Persistent Grade >= 2 sensory neuropathy at enrollment
9. Grade 3 >= hypertension (>= 2 use of antihypertensive drug)
10. Evidence with arterial thromboembolism (Cerebral infarction, Myocardial infarction) or history within 1 year prior to enrollment.
11. Evidence withvenous thromboembolism (deep vein thrombosis, pulmonary embolism) or history within 1 year prior to enrollment.
12. History of GI perforation and/or serious abdominal fistula within 1 year prior to enrollment
13. Cases that the investigator judged as inappropriate as the subject of this clinical study

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Time to failure of strategy (TFS) | 2.5 years

SECONDARY OUTCOMES:
2y Overall Survival rate | 3.5 years
Overall Survival | 3.5years
Progression Free Survival(PFS) | 2.5years
QOL | 2.5years
Biomarker(IMPACT assay Chips, whole blood, tumor tissue, Serum) | 2.5years
  vascular endothelial growth factor(VEGF)-A, VEGFR-2, VEGF-C, platelet derived growth factor(PDGF)-C, Soluble fms-like tyrosine kinase-1, VEGFR-3, Interleukin(IL)-8, Basic Fibroblast Growth Factor(FGFb), placental growth factor(PLGF), E-Selectin, intercellular adhesion molecule(ICAM)-1, neuropilin of Tumor tissue, single nucleotide polymorphism(SNP):VEGFR-1 and VEGF of whole blood DNA, angiotensin(ANG) and Apelin of serum.
Safety(Collection of adverse events) | 2.5years

CONTACTS AND LOCATIONS:
Overall Officials: Masakazu Toi, MD, PhD, Principal Investigator — Kyoto University, Graduate School of Medicine; Shigehira Saji, MD, PhD, Principal Investigator — Fukushima Medical University
Locations (1):
- Japan Breast Cancer Research Group, Chuo-ku, Nihonbashi, Koami-cho, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Deidetified patient data will be made available upon reasonable request.

REFERENCES:
- [Derived] Saji S, Taira N, Kitada M, Takano T, Takada M, Ohtake T, Toyama T, Kikawa Y, Hasegawa Y, Fujisawa T, Kashiwaba M, Ishida T, Nakamura R, Yamamoto Y, Toh U, Iwata H, Masuda N, Morita S, Ohno S, Toi M. Switch maintenance endocrine therapy plus bevacizumab after bevacizumab plus paclitaxel in advanced or metastatic oestrogen receptor-positive, HER2-negative breast cancer (BOOSTER): a randomised, open-label, phase 2 trial. Lancet Oncol. 2022 May;23(5):636-649. doi: 10.1016/S1470-2045(22)00196-6. Epub 2022 Apr 8. PMID 35405087